CLINICAL TRIAL: NCT03404141
Title: Psychological Therapy to Reduce Levels of Stress Among Pregnant Women
Brief Title: Stress Reduction Therapy for Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Borja Romero-Gonzalez, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gestastress
Record Dates: First submitted 2017-12-15; First posted 2018-01-19 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Prenatal Stress
Keywords: Stress; pregnancy; psychological therapy; cortisol
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention administered to the experimental group will be a cognitive-behavior therapy applied by two specifically trained psychologists.
  Due to COVID-19 pandemic, this group will be implemented online using a videocall online platform (from April 2019 to the end of mobility restrictions).
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Control group (Active Comparator): The intervention administered to the control group will consist on a regular parent craft classes offered by the community midwife Due to COVID-19 pandemic, this group will be implemented online using a videocall online platform (from April 2019 to the end of mobility restrictions).
  Interventions: Other: Parent craft

INTERVENTIONS:
Other: Parent craft — Midwife-guided classes for pregnant women about pregnancy and childbirth
  Arms: Control group
Behavioral: Cognitive-Behavioral Therapy — Cognitive-Behavioral Therapy to reduce stress levels among pregnant women
  Arms: Experimental group

SUMMARY:
Prenatal stress is associated with negative outcomes such as postpartum depression, prematurity or neurodevelopmental delays.

The aim of this study is to implement a psychological therapy to reduce stress during pregnancy.

DETAILED DESCRIPTION:
Objective: To assess whether the group of pregnant women have lower levels of stress after attending the psychological therapy than the group attending parent craft classes.

The cognitive-behavioural therapy to reduce stress will be held in 10 sessions (1 per week) as follows:

First session: General information about pregnancy. Pregnant women will describe what can they do to reduce stress levels.

Second session: Breathing techniques and talk about how last week went. Third session: Muscle relaxation and guided imagination techniques Fourth session: Cognitive restructuring. Being able to detect thoughts and feelings Fifth session: Detect cognitive distortions Sixth session: Cognitive restructuring Seventh session: Time management Eighth session: Problems solving Ninth session: Assertively and social skills Tenth session: How to ask for help when needed and learning to say "No".

ELIGIBILITY:
Inclusion Criteria:

* Low risk Pregnant women
* Gestational age between 10-27 weeks
* Proficiency in the Spanish language

Exclusion Criteria:

* Corticoids treatment
* Gestational Diabetes
* Psychological diagnosed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in hair cortisol levels | Baseline, and 3 months
  Change in hair cortisol levels at different time points

SECONDARY OUTCOMES:
Change in Perceived Stress Scale (PSS) | Baseline, and 3 months
  The PSS provides information on the perception of general stress during the preceding month. It consists on 14 items scores on a 5-point Likert scale (0 = never, 1 = almost never, 2 = once in a while, 3 = often, 4 = very often). Scores range from 0-56 (higher scores represent higher levels of stress)
Change in Prenatal Distress Questionnaire (PDQ) | Baseline, and 3 months
  It is a 12-item instrument scored on a 5-point Likert scale from 0 (none at all) to 4 (extremely) to assess specific worries and concerns pregnant women experience regarding medical problems, physical symptoms, body changes, labor, childbirth, relationships, and the baby's health. Scores range from 0-48 (higher scores represent higher levels of pregnancy specific-stress)
Change in Symptoms Checklist 90 Revised (SCL-90-R) | Baseline, and 3 months
  This is a 90-item scale scored using a 5-point Likert scale from 0 (never) to 4 (extremely). This instrument is used to assess 9 dimensions: Somatization, Obsession-compulsion, Interpersonal sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation, and Psychoticism. The scale also has 7 extra items distributed among 3 global indexes of distress: the GSI, which measures overall psychological distress; the PSDI, which is used to measure the intensity of symptoms; and Positive Symptom Total, used to measure the number of self-reported symptoms. Using the author´s instructions, the scores are transformed to percentiles (0-100). Percentiles ≥ 70 represent clinical symptoms in any of the subscale of this instrument.
Change in Connor-Davidson Resilience Scale (CD-RISC) | Baseline, and 3 months
  It consists of 25 items evaluated on a 5-point Likert scale ranging from 0-4: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4) - these ratings result in a number between 0-100, and higher scores indicate higher resilience.

OTHER OUTCOMES:
Infant neurodevelopment | 6 months of age
  Infant neurodevelopment at 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Borja Romero, Principal Investigator — Universidad de Granada
Locations (1):
- Granada, Churriana de la Vega, Granada, Spain

REFERENCES:
- [Derived] Romero-Gonzalez B, Puertas-Gonzalez JA, Strivens-Vilchez H, Gonzalez-Perez R, Peralta-Ramirez MI. Effects of cognitive-behavioural therapy for stress management on stress and hair cortisol levels in pregnant women: A randomised controlled trial. J Psychosom Res. 2020 Aug;135:110162. doi: 10.1016/j.jpsychores.2020.110162. Epub 2020 May 26. PMID 32485622